CLINICAL TRIAL: NCT02960477
Title: Effectiveness of Pain Neuroscience Education vs Biomedical Education for Patients Undergoing Surgery for Shoulder Pain: Protocol for a Randomized Controlled Trial
Brief Title: Effectiveness of Pain Neuroscience Education vs Biomedical Education for Patients Undergoing Surgery for Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Malaga
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2017-11

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain; Shoulder surgery; Pain neuroscience education; Chronic pain
MeSH Terms: conditions — Shoulder Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience education (Experimental): A PNE session covers the neurobiology, neurophysiology and processing of pain. Topics addressed during the educational sessions will include the characteristics of acute versus chronic pain; how pain becomes chronic (plasticity of the nervous system, modulation, modification, central sensitization, etc.); potential sustaining factors of central sensitization like emotions, stress, pain cognitions, and pain behaviour; the decision to have shoulder surgery; surgical experiences and environmental issues' effects on nerve sensitivity; recovery after shoulder surgery; scientific evidence for the PNE content; and the opportunity to reflect and write questions to ask the surgeon prior to surgery.
  Interventions: Other: Pain Neuroscience education
- Biomedical Education (Active Comparator): A biomedical session covers the normal course of shoulder pain; anatomy, physiology and biomechanics of the shoulder; the expected course of postoperative shoulder pain; and the importance of self-care. Also, professional and leisure time activities will be discussed. Ergonomic advices will be given: e.g. how is the best way to catch a container, how I should move my shoulder in this sport/activity, what is a good work posture? The content of the biomedical education will be biomedically-/biomechanically-focussed.
  Interventions: Other: Biomedical Education

INTERVENTIONS:
Other: Pain Neuroscience education — A PNE session covers the neurobiology, neurophysiology and processing of pain.
  Arms: Pain Neuroscience education
Other: Biomedical Education — A biomedical session covers the normal course of shoulder pain, anatomy, physiology and biomechanics of the shoulder, the expected course of postoperative shoulder pain, and the importance of self-care.
  Arms: Biomedical Education

SUMMARY:
BACKGROUND Shoulder pain is the third most common musculoskeletal disorder observed in primary care consultations after low back and neck pain. In the absence of successful outcome following a conservative intervention, shoulder surgery is the most common procedure conduct for a multitude of surgical indications, including rotator cuff tears, instability and stiffness. However, 22% of patients develop chronic shoulder pain (CSP) following shoulder surgery . The consequences of chronic or persistent postsurgical pain result in high socio-economic burden, not only in terms of suffering and reduced quality of life for the individual, but also, with considered the subsequent costs to healthcare and social services.

Pain neuroscience education (PNE) has been shown as an effective therapeutic strategy for increasing knowledge and understanding about neurobiology, neurophysiology and processing pain, changing pain beliefs, improving patient's skills and encouraging to do physical and social activities in different chronic pain conditions.

The primary aim of this study will be to evaluate whether perioperative PNE is more effective than classical biomedical education in reducing pain and disability in patients undergoing shoulder surgery. The secondary aim will be to analyse whether perioperative PNE is more effective than classical biomedical education in reducing postoperative healthcare costs and improving surgical experience in patients undergoing shoulder surgery .

DETAILED DESCRIPTION:
The present study will be a 6-month randomized controlled trial that will be carried out between March 2017 and Aug 2017 in a regional hospital (secondary care setting ) of the province of Malaga, Spain. Participants scheduled for shoulder surgery and those that fulfil inclusion criteria will be asked for participating in this study. The outcomes will be assessed at baseline (in the week preceding surgery) and at 3 follow-ups times (1 week, 1 month and 6 months' post-surgery t1-t4 ).

All patients scheduled for shoulder surgery in the participating hospital and meeting the age criteria will be contacted by telephone and interviewed after having given consent. The initial telephone interview serves to provide a verbal description of the project and to screen potential study participants for in- and exclusion criteria (see above). People deemed likely to be eligible and willing to participate in the study will be scheduled for baseline assessments in the week before surgery. Furthermore, they will receive written information about the study via mail or e-mail. Prior to undertaking the baseline assessments, they will have the opportunity to ask questions and will be asked to provide written informed consent. Anonymized age, gender and visual analogue scale- verbal numerical rating scale (VAS-VNRS) for pain will be collected for those participants who decline to take part in the project, to assess the external validity of the recruited sample of participants.

Participants are not expected to start new treatments or medication other than their usual pre- and postoperative care 3 weeks prior to and during study participation. Participants will then complete several questionnaires at baseline, 1 week, 1 month and 6 months' post-intervention apart from biomedical education or PNE intervention. Retention of participants will be encouraged by researchers providing written feedback to all participants about the results of the "health screenings", maintaining the interest in the study through materials and mailings sent to participants during all the process and using reminders of the upcoming data collection. Participant data files will be stored in numerical order and in a secure and accessible place and manner. Participant files will be maintained in storage for a period of 3 years after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for shoulder surgery, willing to participate (including willingness to comply with the predetermined follow-ups).
2. Participants scheduled for shoulder surgery due to partial or full thickness rotator cuff tear, tendon biceps tears, impingement syndrome, rotator cuff tendinopathy, adhesive capsulitis, rotator cuff tendinosis and labral pathologies will be included in this study. Diagnosis will be based on surgeon criteria and confirmed by MRI or US .
3. Men / women aged between 18 and 70 years.

Exclusion Criteria:

1. Chronic illness characterized by chronic pain (e.g. rheumatoid arthritis, fibromyalgia, chronic fatigue syndrome, scleroderma) or any other rheumatoid, endocrinological, neurological or psychiatric disorder.
2. Patients with evidence of advanced osteoarthritis of the glenohumeral joint and inflammatory arthropathy .
3. Shoulder pain considered to be originated from the cervical region and other traumas or if there is osteoporosis, haemophilia and / or cancer.
4. Participants receiving shoulder surgery before the beginning of the study.
5. Inability to provide informed consent and/or complete written questionnaires.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
"Change from Baseline pain and function at 6 months" | 6 months
  This outcome will be measured with the shoulder pain and disability index (SPADI)

SECONDARY OUTCOMES:
"Change from Baseline patient's expectations of surgical experience at 6 months" | 6 months
  To assess surgical experience, patients will be asked to indicate the level of agreement (on a numerical rating scale from 1 "minimal" to 10 "maximal agreement") with statements about their shoulder surgery/education experience: "I am glad I underwent surgery for my shoulder."; "I was fully prepared (physically, emotionally, and psychologically) for the surgery."; "The preoperative education I received prepared me well for the surgery."; "Knowing what I know now, I would do this again given the same choices." and "The surgery met my expectations.".
"Change from Baseline postoperative healthcare costs at 6 months" | 6 months
  Postoperative healthcare costs include the number of days spent in hospital following surgery, medical tests related to postoperative surgery and any kind of postoperative treatments (e.g. pain killers, physiotherapy, psychotherapy, osteopathy).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Luque Suarez, PhD, Principal Investigator — University of Malaga

IPD SHARING:
Plan to Share IPD: No